CLINICAL TRIAL: NCT06201000
Title: Effect of Genetic Polymorphisms on the Clinical Response to Sodium-glucose Cotransporter 2 (SGLT2) Inhibitors in Prevention of Cardiac Remodeling and Fibrosis in Heart Failure Patients
Brief Title: Effect of Genetic Polymorphisms on the Clinical Response to SGLT2 Inhibitors in Heart Failure Patients
Status: Recruiting | Type: Observational
Sponsor: October 6 University (Other)
Collaborators: University of Florida (Other); National Heart Institute, Egypt (Other Government); Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Essam, Assistant Lecturer in Clinical Pharmacy Department, October 6 University
Other Study IDs: IHC00068
Record Dates: First submitted 2023-12-27; First posted 2024-01-11 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Genetic Polymorphisms; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Heart Failure Patients with reduced or preserved Ejection Fraction: Patients with reduced or preserved ejection fraction that have received the Guided Therapy (β-blockers, Diuretics, Angiotensin-converting enzyme (ACE) inhibitors or Angiotensin receptor blockers (ARBs) or Angiotensin Receptor-Neprilysin Inhibitor (ARNi) and Mineralocorticoid receptor antagonists (MRAs) then Sodium-glucose cotransporter-2 inhibitors (SGLT-2i) (10 mg of dapagliflozin or empagliflozin) will be added at the study entry.
  Interventions: Drug: SGLT2 inhibitors (Dapagliflozin and Empagliflozin)

INTERVENTIONS:
Drug: SGLT2 inhibitors (Dapagliflozin and Empagliflozin) — 10 mg of dapagliflozin or empagliflozin
  Other Names: Forxiga; Jardiance

SUMMARY:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors have shown further reductions in heart failure hospitalization, cardiovascular events, and mortality, especially for heart failure patients.

The SGLT2 gene, also known as SLC5A2 (solute carrier family 5 member 2), is located on chromosome 16 and is responsible for encoding SGLT2.

Several SLC5A2 mutations alter SGLT2 expression, membrane location, or transporter function.

Several common genetic variations were found in the SLC5A2 gene that may affect the response to treatment with SGLT2 inhibitors.

DETAILED DESCRIPTION:
Sodium-glucose cotransporter-2 inhibitors (SGLT-2i), which were first investigated and licensed for the treatment of diabetes, are now emerging as a promising class of drugs for the treatment of heart failure (HF), even in people without diabetes.

Significant reductions in worsening heart failure or cardiovascular death were shown under treatment with dapagliflozin and empagliflozin in the trials of patients with heart failure.

Several common genetic variations were found in the SLC5A2 gene that may affect the response to treatment with SGLT2 inhibitors.

The most recent SLC5A2 Single Nucleotide Polymorphisms (SNPs) that reduce the risk of heart failure included two intronic SLC5A2 SNPs, s9934336, and rs3116150, both associated with the expression levels of the transporter.

This study aims to detect the association between SLC5A2 single nucleotide polymorphisms and variability in response to SGLT2 Inhibitors as well as the association between cardiac biomarkers and non-coding RNA in patients with Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients NYHA class II to III.
* Heart failure patients with reduced left ventricular ejection fraction (LVEF) < 45% or with preserved left ventricular ejection fraction (LVEF) > 45%
* Patients who will be candidate for add-on treatment with SGLT2.
* Patients who will be able to sign informed consent to participate in the study.

Exclusion Criteria:

* Contraindications to SGLT2.
* Significant coronary artery diseases (CAD), coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), or valve surgery within 3 months.
* Pregnant or breastfeeding women.
* Patients with estimated glomerular filtration rates less than 30 mL/min/1.73 m2, as determined using the CKD-EPI equation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of established Heart failure with reduced ejection fraction (HFrEF) or Heart failure with preserved ejection fraction (HFpEF) and New York Heart Association (NYHA) functional classes II-III, who will be candidates for add-on treatment with SGLT2i.
Sampling Method: Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Median / Mean of Left Ventricular Ejection Fraction (LVEF) among studied genetic polymorphisms | 6 months
  Change in median / mean of Left Ventricular Ejection Fraction (LVEF) before and after drug administration
Median / Mean of Left Ventricular End Systolic Volumes among studied genetic polymorphisms | 6 months
  Change in median / mean of Left Ventricular End Systolic Volume (LVESV)
Median / Mean of Left Ventricular End Diastolic Volumes among studied genetic polymorphisms | 6 months
  Change in median / mean of Left Ventricular End Diastolic Volume (LVEDV) before and after drug administration

SECONDARY OUTCOMES:
Median / Mean of quality of life measure {Kansas City Cardiomyopathy Questionnaire (KCCQ-12)} among studied genetic polymorphisms | 6 months
  Change in median / mean of Kansas City Cardiomyopathy Questionnaire (KCCQ-12) before and after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Rania Sarhan, PhD, Study Director — Beni-Suef University; Neven Sarhan, PhD, Study Director — Misr International University; Bassem Zarif, MD, Study Director — National Heart Institute; Julio Duarte, PhD, Study Chair — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States